CLINICAL TRIAL: NCT05065151
Title: Understanding Motivation in Parkinson's Patients Through Neurophysiology
Acronym: MPPN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Yale University (Other); Rune Labs (Unknown); University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20-31239
Record Dates: First submitted 2021-09-17; First posted 2021-10-01 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease; Deep Brain Stimulation; Motivation
Keywords: Parkinson's; Medtronic; Percept; DBS; Deep Brain Stimulation; Parkinson's Disease; Parkinson Disease; PD; Reward-based decision making; Task
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Within subject crossover counterbalanced study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Stimulation (Experimental): Patients will be getting standard clinically acceptable stimulation within already safety validated stimulation ranges through their Medtronic Percept device.
  Interventions: Other: Stimulation on; Behavioral: Decision Making Task
- No Stimulation (Experimental): Patients will have stimulation turned off through their Medtronic Percept device.
  Interventions: Other: Stimulation off; Behavioral: Decision Making Task

INTERVENTIONS:
Other: Stimulation on — Stimulation from Percept DBS will be on while the patient is playing a decision-making game on a computer-based application.
  Other Names: Medtronic Percept
  Arms: Stimulation
Other: Stimulation off — Stimulation from Percept DBS will be off while the patient is playing a decision-making game on a computer-based application.
  Other Names: Medtronic Percept
  Arms: No Stimulation
Behavioral: Decision Making Task — Patients will be playing a decision making task through a computer-based application.

SUMMARY:
The study aims to better understand motivation and value-based decision-making in Parkinson's patients through neurophysiology using Medtronic's Percept DBS device. By combining behavioral tasks with neural recordings, the study seeks to uncover how DBS affects motivation, particularly in relation to effort, reward, and timing.

DETAILED DESCRIPTION:
Participants will perform reward-based decision-making tasks designed to assess both self-benefitting and prosocial motivation. The tasks will evaluate how effort and reward influence decision-making, as well as how proximity to a deadline impacts choices. These tasks will be conducted in both clinic and home settings.

Throughout the study, participants will remain on their regular dopaminergic medications. Each participant will complete sessions under two stimulation conditions: their usual DBS settings and with DBS turned off. Neural activity will be recorded using the Percept device, which enables real-time and chronic at-home data streaming. Additionally, participants will wear a device that captures movement, sleep, heart rate variability, and self-reported measures.

The primary outcomes are behavioral: changes in reaction time, acceptance rate, and success rate across different DBS conditions. The secondary outcomes focus on identifying neural oscillatory biomarkers time-locked to specific decision-making events. By linking brain activity to motivational behavior, this study aims to advance our understanding of non-motor symptoms in PD and inform the development of adaptive DBS algorithms targeting these symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Has Parkinson's Disease or Dystonia
* Has Medtronic Percept or RC+S DBS device implanted in either GPI or STN
* Has DBS device implanted either bilaterally or unilaterally
* Male or female
* More than 1 month post-DBS surgery

Exclusion Criteria:

* Severe cognitive impairments
* Has MOCA score below 20
* Pregnancy
* Age less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-10-30 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Percent of Risky Decisions made with Percept DBS stimulation on for Parkinson's Disease Patients | The values will be collected starting from admission in clinic and the at-home paradigm. Data collection and analysis of said values can take up to three years
  Patients' responses on the tablet will be recorded in-clinic and at home. The investigators will tally their choices from the value-based decision making game (risky versus safe decisions) and report an average of risky responses.
Percent of Risky Decisions made with Percept DBS stimulation off for Parkinson's Disease Patients | The values will be collected starting from admission in clinic and the at-home paradigm. Data collection and analysis of said values can take up to three years
  Patients' responses on the tablet will be recorded in-clinic and at home. The investigators will tally their choices from the value-based decision making game (risky versus safe decisions) and report an average of risky responses.
Reaction Time During Decision-Making Task | The values will be collected starting from admission in clinic. Data collection and analysis of said values can take up to three years.
  The investigators will measure the time it takes for patients to make each decision on the value-based decision-making task in the clinic.
Task Success Rate | The values will be collected starting from admission in clinic. Data collection and analysis of said values can take up to three years.
  The investigators will calculate the percentage of trials in which patients complete the task successfully according to predefined task performance criteria.
Acceptance Rate of Risky Versus Safe Options | The values will be collected starting from admission in clinic. Data collection and analysis of said values can take up to three years.
  The proportion of trials where patients accept risky versus safe options will be calculated and compared across stimulation ON and OFF conditions.
Force Exertion During Motor Responses | The values will be collected starting from admission in clinic. Data collection and analysis of said values can take up to three years.
  Force data will be recorded during motor responses to evaluate physical engagement and motor control during task performance.
Low frequency local field potentials | The values will be collected starting from admission in clinic. Data collection and analysis of said values can take up to three years.
  Local field potentials (LFPs) will be recorded from the implanted Percept device to evaluate neural activity during decision making under different stimulation conditions. Low frequency power will be calculated during specific time intervals during the task. Cardiac artifact will be removed with electrocardiogram (ECG) measurements recorded during the same task.
Electroencephalogram (EEG) theta band power | The values will be collected starting from admission in clinic. Data collection and analysis of said values can take up to three years.
  Scalp EEG will be recorded concurrently with task performance to assess cortical activity patterns during decision-making. Average theta band power will be calculated in specific time intervals during the task.
Electroencephalogram (EEG) beta band power | The values will be collected starting from admission in clinic. Data collection and analysis of said values can take up to three years.
  Scalp EEG will be recorded concurrently with task performance to assess cortical activity patterns during decision-making. Average beta band power will be calculated in specific time intervals during the task.
Electroencephalogram (EEG) gamma band power | The values will be collected starting from admission in clinic. Data collection and analysis of said values can take up to three years.
  Scalp EEG will be recorded concurrently with task performance to assess cortical activity patterns during decision-making. Average gamma band power will be calculated in specific time intervals during the task.
Electroencephalogram (EEG) alpha band power | The values will be collected starting from admission in clinic. Data collection and analysis of said values can take up to three years.
  Scalp EEG will be recorded concurrently with task performance to assess cortical activity patterns during decision-making. Average alpha band power will be calculated in specific time intervals during the task.

SECONDARY OUTCOMES:
Interaction Between Neural Low Frequency Power in the LFP with Reaction Time (seconds) | Analysis will occur continuously throughout the study period (up to three years) based on collected behavioral and neural data.
  We will assess the effect of reaction time on low frequency power in the LFP data (theta, alpha, beta power) recorded from the Percept device with statistical modeling.
Interaction Between Neural Low Frequency Power in the LFP with Success Rate (percentage) | Analysis will occur continuously throughout the study period (up to three years) based on collected behavioral and neural data.
  We will assess the effect of success rate on low frequency power in the LFP data (theta, alpha, beta power) recorded from the Percept device with statistical modeling.
Interaction Between Neural Low Frequency Power in the LFP with Force Exerted (arbitrary units) | Analysis will occur continuously throughout the study period (up to three years) based on collected behavioral and neural data.
  We will assess the effect of force exerted on low frequency power in the LFP data (theta, alpha, beta power) recorded from the Percept device with statistical modeling.
Interaction Between Neural Low Frequency Power in the EEG with Reaction Time (seconds) | Analysis will occur continuously throughout the study period (up to three years) based on collected behavioral and neural data.
  We will assess the effect of reaction time on low frequency power in the EEG data (theta, alpha, beta power) recorded from the Percept device with statistical modeling.
Interaction Between Neural Low Frequency Power in the EEG with Success Rate (percentage) | Analysis will occur continuously throughout the study period (up to three years) based on collected behavioral and neural data.
  We will assess the effect of success rate on low frequency power in the EEG data (theta, alpha, beta power) recorded from the Percept device with statistical modeling.
Interaction Between Neural Low Frequency Power in the EEG with Force Exerted (arbitrary units) | Analysis will occur continuously throughout the study period (up to three years) based on collected behavioral and neural data.
  We will assess the effect of force exerted on low frequency power in the EEG data (theta, alpha, beta power) recorded from the Percept device with statistical modeling.

CONTACTS AND LOCATIONS:
Overall Officials: Simon J Little, MBBS, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Future data sharing will be covered by UCSF data sharing compliance rules.

REFERENCES:
- [Background] Rutledge RB, Skandali N, Dayan P, Dolan RJ. A computational and neural model of momentary subjective well-being. Proc Natl Acad Sci U S A. 2014 Aug 19;111(33):12252-7. doi: 10.1073/pnas.1407535111. Epub 2014 Aug 4. PMID 25092308
- [Background] Rutledge RB, Skandali N, Dayan P, Dolan RJ. Dopaminergic Modulation of Decision Making and Subjective Well-Being. J Neurosci. 2015 Jul 8;35(27):9811-22. doi: 10.1523/JNEUROSCI.0702-15.2015. PMID 26156984
- [Background] Eldar E, Rutledge RB, Dolan RJ, Niv Y. Mood as Representation of Momentum. Trends Cogn Sci. 2016 Jan;20(1):15-24. doi: 10.1016/j.tics.2015.07.010. Epub 2015 Nov 3. PMID 26545853
- [Background] Blain B, Rutledge RB. Momentary subjective well-being depends on learning and not reward. Elife. 2020 Nov 17;9:e57977. doi: 10.7554/eLife.57977. PMID 33200989
- [Background] Talbot J, Cutler J, Tamm M, Little SJ, Harmer CJ, Husain M, Lockwood PL, Apps MAJ. Dopamine boosts motivation for prosocial effort in Parkinson's disease. J Neurosci. 2025 Jan 2:e1593242024. doi: 10.1523/JNEUROSCI.1593-24.2024. Online ahead of print. PMID 39746820
- [Background] Pisauro MA, Pollicino D, Fisher L, Apps MAJ. Neural and computational mechanisms of effort under the pressure of a deadline. bioRxiv. 2024. doi:10.1101/2024.04.17.589910.